CLINICAL TRIAL: NCT07137247
Title: Immune Dynamics in the Natural History of Chronic HBV Infection
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-216
Record Dates: First submitted 2025-06-19; First posted 2025-08-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: HBV (Hepatitis B Virus); HBV Infection; Chronic Hep B
Keywords: HBV; Chronic Hep B; HBV infection
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic hepatitis B virus (HBV) infection: Patients with chronic HBV infection who are untreated and aged 1-80 years. Follow-ups will be conducted every six months, with a minimum of six visit points.
  Interventions: Procedure: Venipuncture

INTERVENTIONS:
Procedure: Venipuncture — For adults (including those who are 18 years old): During the routine follow-up visits, an extra 30 milliliters of peripheral blood will be drawn.
  For minors (under 18 years old): During the routine follow-up visits, an extra 6 milliliters of peripheral blood will be drawn.
  Follow-ups will be conducted every six months, with a minimum of six visit points.

SUMMARY:
The purpose of this observational study is to follow up on chronic HBV-infected patients over a long period of time to understand the changes in the immune status as age increases and the natural history of chronic HBV infection progresses. The main questions it aims to answer are:

* Does the natural history of chronic HBV infection progress with changes in HBV-specific immunity?
* What is the role of age in the natural history of chronic HBV infection?

Patients with chronic HBV infection who are untreated and aged 1-80 years will be followed up every six months. During each follow-up, HBV-related serological and virological indicators will be tested. Peripheral blood samples will also be collected to test HBV-specific immunity and the immune environment.

DETAILED DESCRIPTION:
Research Objectives This study aims to investigate the mechanisms underlying the changes and potential deficiencies in humoral and cellular immunity caused by chronic HBV infection through the analysis of clinical samples from patients with hepatitis B. Clinical Investigator will compare the differences in the generation, proliferation, and survival of immune cells among patients with chronic hepatitis B at different immune status stages and explore the role and mechanisms of these differences in anti-HBV immunity. Additionally, clinical Investigator will evaluate their potential impact on the functional cure of hepatitis B.

Study Design As this is an observational study, patients will not be required to undergo additional visits or laboratory tests beyond routine clinical practice. The treatment plan will be determined by the physician according to the instructions and local guidelines. Researchers will review the patient's medical history and laboratory reports to determine eligibility based on inclusion and exclusion criteria. Patients must sign the latest informed consent form approved by the ethics committee before data collection. The frequency and timing of visits will be decided by the physician according to local routine practices. In line with routine clinical practice, follow-ups will be conducted every six months. In this study, laboratory and clinical assessment data will be collected at baseline and every six months. Each participant will be assigned a unique identification number (e.g., HBV1, HBV2), which will be used for all study documents (such as case report forms and clinical records). Participants who meet all inclusion and exclusion criteria and sign the informed consent form will be enrolled in the study. In accordance with data privacy regulations, the use of unique identification numbers is permitted as long as they do not contain combinations of information that can identify participants (for example, the use of participants' initials and date of birth together is not allowed). Participants who withdraw from the study midway will be considered dropouts. When a participant drops out, researchers should try to contact the participant to complete the relevant assessments and fill out the study summary page. Data for this study will be obtained by extracting the participants' routine clinical medical records. Researchers are required to fill out the electronic case report form (eCRF) based on the information in the patient's medical records.

Data Collection Procedures

Baseline Period :

Demographic Data: Record date of birth, gender, and initials. Medical History: Record etiology, current illness history, past medical history, and medication history.

Physical Examination: Check vital signs, height, and weight; observe for the presence of spider angiomas or palmar erythema, dull complexion, jaundice of skin and sclera, hepatic pain, and splenomegaly.

Blood Draw: In addition to routine blood tests, an additional 30ml of blood will be drawn from adults (6ml for minors) for basic experiments and flow cytometry to detect changes in the phenotype and function of immune cells (T cells, B cells, monocytes, etc.) in patients with chronic HBV infection, as well as the frequency of HBV-specific T cells and B cells in patients at different clinical stages, in order to identify biomarkers associated with the prognosis of HBV infection.

Routine Treatment Period :

Medical History: Record current illness history, past medical history, and medication history.

Physical Examination: Check vital signs, height, and weight; observe for the presence of spider angiomas or palmar erythema, dull complexion, jaundice of skin and sclera, hepatic pain, and splenomegaly.

Blood Draw: Blood will be drawn once at each of the six routine treatment visits. In addition to routine blood tests, an additional 30ml of blood will be drawn from adults (6ml for minors) for basic experiments and flow cytometry to detect changes in the phenotype and function of immune cells in patients with chronic HBV infection, as well as the frequency of HBV-specific T cells and B cells in patients at different clinical stages, in order to identify biomarkers associated with the prognosis of HBV infection.

The efficacy observation includes: quantitative hepatitis B virus DNA, hepatitis B surface antigen, hepatitis B e antigen, and hepatitis B e antibody. Depending on the needs of routine clinical diagnosis and treatment, additional tests such as imported quantitative hepatitis B virus DNA (HBV DNA cobas), alpha-fetoprotein, hepatitis B core antibody, and liver stiffness scan may be performed.If patients undergo additional tests for quantitative hepatitis B virus DNA (HBV DNA cobas), alpha-fetoprotein, hepatitis B core antibody, and liver stiffness scan as part of routine clinical care, the study will also collect these data.

Sample Collection:

Adult Participants (including those aged 18 years): Blood samples will be collected once at the baseline visit and at each of the six routine treatment visits. An additional 30ml of blood will be drawn at each visit, specifically in three sodium heparin anticoagulant tubes (10ml per tube).

Minor Participants: Blood samples will be collected once at the baseline visit and at each of the six routine treatment visits. An additional 6ml of blood will be drawn at each visit, specifically in one 6ml sodium heparin anticoagulant tube.

Safety Monitoring, Reporting, and Medical Management:

Adverse Event (AE) Definition: An adverse event is any untoward medical occurrence in a patient or participant after the administration of a drug, which does not necessarily have a causal relationship with the treatment. Adverse events can be any adverse signs (including abnormal laboratory findings), symptoms, or diseases related to the use of the study drug in terms of timing, regardless of whether they are considered to have a causal relationship with the study drug. Adverse events include serious adverse events (Serious Adverse Event, SAE) and non-serious adverse events.

SAE Definition: An SAE is a medical event that occurs during a clinical study and requires hospitalization or prolongation of hospital stay, causes disability, affects the ability to work, is life-threatening or fatal, or leads to congenital anomalies. It includes the following medical events:

Events leading to death; Life-threatening events (defined as events where the participant is at immediate risk of death at the time of the event); Events requiring hospitalization or prolongation of hospital stay; Events that can cause permanent or severe disability/functional impairment/loss of ability to work; Congenital abnormalities or birth defects; Other important medical events (defined as events that endanger the participant or require intervention to prevent any of the above situations from occurring).

AE Collection, Reporting, and Management:

All AEs related to the study protocol procedures that occur after signing the informed consent form and before taking the study drug must be recorded in the eCRF. The record of AEs should include: a description of the AE and all related symptoms, time of occurrence, severity, duration, relationship to the study drug, measures taken, and final outcome and resolution. The recording of AEs must use medical terminology. If the participant's symptoms and signs can be attributed to a common etiology, a diagnosis should be recorded whenever possible. Except for disease progression-related indicators, all clinical events and laboratory adverse reactions of clinical significance can be managed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse reactions caused by treatment will be recorded by the researcher.

SAE Collection and Reporting:

All SAEs that occur from the time the participant signs the informed consent form to the end of the 96-week post-treatment observation period must be reported using an SAE report form, regardless of the cause or relationship to the drug. If an SAE occurs, the researcher should immediately take appropriate therapeutic measures for the participant to ensure their safety and report to the drug registration applicant, the National Medical Products Administration, the Provincial Food and Drug Administration, the corresponding clinical research center ethics committee, and the Medical Administration Department of the National Health Commission within 24 hours. The report should also be promptly submitted to the ethics committee of the lead unit. The initial report should include the following information whenever possible: source of the report, name of the study drug, name of the serious adverse event, time of occurrence, severity, duration, relationship to the study drug, measures taken, and outcome.

AE Severity Assessment Criteria:

Researchers will assess the severity based on the five-level grading criteria established by the NCI CTCAE version 5.0:

Grade 1: Mild; asymptomatic or with only slight signs; for clinical or diagnostic observation only, without the need for medical intervention; Grade 2: Moderate; limitation of daily living activities appropriate for age (such as cooking, shopping, making phone calls); Grade 3: Severe or of significant medical importance but not immediately life-threatening; resulting in hospitalization or prolongation of hospital stay; disability; limitation of activities of daily living (activities of daily living refer to bathing, dressing, undressing, eating, toileting, taking medication, etc., but not bedridden); Grade 4: Life-threatening, requiring urgent treatment; Grade 5: Related to the Death 6. Statistical Analysis Sample Size Determination: This study is exploratory in nature and does not focus on the impact of sample size on clinical endpoints. Research Objectives This study aims to investigate the mechanisms underlying the changes and potential deficiencies in humoral and cellular immunity caused by chronic HBV infection through the analysis of clinical samples from patients with hepatitis B. Clinical Investigator will compare the differences in the generation, proliferation, and survival of immune cells among patients with chronic hepatitis B at different immune status stages and explore the role and mechanisms of these differences in anti-HBV immunity. Additionally, clinical Investigator will evaluate their potential impact on the functional cure of hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-80 years, either male or female.
* Patients diagnosed with chronic hepatitis B virus infection in accordance with the "Guidelines for the Prevention and Treatment of Chronic Hepatitis B" (2019 edition).
* No antiviral treatment (including nucleoside analogs and interferons, etc.) within the past six months.

Exclusion Criteria:

• Concurrent Infections and Liver Diseases: Exclusion of patients with concurrent HCV or HIV infection, alcoholic fatty liver disease, non-alcoholic fatty liver disease, autoimmune liver diseases.

• Immune and Coagulation System Disorders: Exclusion of patients with immune system diseases such as hyperthyroidism, coagulation system disorders such as diabetes mellitus or idiopathic thrombocytopenic purpura.

* Severe Underlying Diseases. Exclusion of patients with severe underlying diseases that affect the body's immune status.
* Other Unsuitable Conditions:

Exclusion of patients whom the investigator deems to have other conditions that make them unsuitable for enrollment.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of chronic hepatitis B patients who have not received antiviral therapy within the past six months.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2040-12-01 (Estimated); Study Completion 2041-12-01 (Estimated)

PRIMARY OUTCOMES:
In accordance with the 2018 AASLD Hepatitis B guidelines, the natural history of HBV is staged based on the laboratory test results (HBV serological markers, viral load, and liver function) and imaging findings of the enrolled patients. | over a follow-up period of 5 years
  Enrolled patients will undergo examinations of HBV serological markers, viral load, liver function, liver ultrasound, and liver fibrosis every six months. Subsequently, based on the 2018 AASLD Hepatitis B guidelines , patients will be staged to observe whether there are changes in the natural history of hepatitis B.

SECONDARY OUTCOMES:
The HBV-specific immune response levels will be measured using the immune cells of the enrolled patients | over a follow-up period of five years
  During the biannual follow-up visits, blood samples from the enrolled patients will be used to detect the levels of HBV-specific immunity and other laboratory indicators after restimulation with HBV peptide pools

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No